CLINICAL TRIAL: NCT06881550
Title: A Single-center, Real-world Study of Shenbailing Granules in Patients After Breast Cancer Surgery
Brief Title: Real-world Study on Shenbailing Granules for Improving Qi and Blood Deficiency in Patients After Breast Cancer Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Caigang Liu (Other)
Responsible Party: Sponsor-Investigator, Caigang Liu, Postdoctoral, Chief Physician, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBL-RWS
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Normal postoperative recovery without Shenbailing granules
- TCM (Experimental): Adjuvant therapy with Shenbailing granules, starting from 1 day after surgery
  Interventions: Drug: Shenbailing

INTERVENTIONS:
Drug: Shenbailing — Adjuvant therapy with Shenbailing granules, starting from 1 day after surgery.
  Arms: TCM

SUMMARY:
This study aims to explore the clinical efficacy of Shenbailing granules in improving quality of life and reducing cancer-related fatigue in a real-world setting, with the goal of providing clinical evidence for the use of Shenbailing granules in alleviating cancer-related fatigue among post-breast cancer surgery patients.

DETAILED DESCRIPTION:
This study plans to enroll patients who have undergone breast cancer surgery. The experimental group will receive Shenbailing granule therapy, with the primary objective of exploring the improvement of postoperative cancer-related fatigue and quality of life in breast cancer patients treated with Shenbailing granules. Patients will enter the real-world study phase immediately after surgery.

Experimental group: Adjuvant therapy with Shenbailing granules, starting from 1 day after surgery; Control group: Normal postoperative recovery without medication.

After confirming the surgery date, patients' quality of life, cancer-related fatigue, and breast cancer patient-reported outcome scales will be collected preoperatively, 1 day, 7 days, 14 days, and 28 days postoperatively to evaluate their quality of life and cancer-related fatigue. If patients are not tolerant to the medication, they will stop taking it.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following enrollment criteria to be enrolled in this trial:

1. be 18-75 years of age (both 18 and 75);
2. female;
3. all patients have histologically confirmed breast cancer;
4. expected to receive surgical treatment;
5. expected survival of ≥ 1 year;
6. the level of function of vital organs must meet the following requirements:

   1. Bone marrow function Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L; Platelets ≥ 100 x 10^9/L; Hemoglobin ≥ 90 g/L;
   2. Liver and kidney function Albumin level ≥ 3.0 g/dL; Total bilirubin ≤ 1.5 x upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; Alkaline phosphatase ≤ 2.5 x ULN; Urea nitrogen and serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 60 mL/min (calculated according to the Cockcroft-Gault formula);
   3. Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN;
   4. Echocardiogram (ECHO) showing cardiac left ventricular ejection fraction (LVEF) ≥ 50%;

8. voluntarily accept the treatment and sign the informed consent form, have understood the purpose of this study and the experimental steps, good compliance, and comply with the relevant requirements of this trial protocol.

Exclusion Criteria:

1. intolerance to or poor compliance with herbal medicines;
2. inability to swallow, chronic diarrhea and intestinal obstruction, and the presence of multiple factors affecting the administration and absorption of medications;
3. severe cardiac, hepatic, renal and other vital organ insufficiency;
4. combination of serious complications, active infection, persistent fever, serious bleeding tendency, hematopoietic function abnormality;
5. a known history of allergy to the drug components of this regimen;
6. have a history of immunodeficiency, including testing positive for HIV, HCV, active viral hepatitis B, or suffering from other acquired, congenital immunodeficiency diseases, or have a history of organ transplantation
7. a history of any cardiac disease, including (1) arrhythmia requiring medication or of clinical significance, (2) myocardial infarction, (3) heart failure, (4) any other cardiac disease judged by the investigator to be inappropriate for participation in the study, etc;
8. pregnant or lactating female patients, female patients of childbearing potential with a positive baseline pregnancy test or female patients of childbearing potential who are unwilling to use effective contraception throughout the trial period;
9. in the judgment of the investigator, have a serious concomitant medical condition that jeopardizes the patient's safety, or interferes with the patient's ability to complete the study (including, but not limited to, severe hypertension that cannot be controlled by medication, severe diabetes mellitus, active infection, etc.)
10. is unconscious, non-verbal or non-reading, unable to communicate normally, and unable to cooperate in completing the questionnaire assessment;
11. a previous history of a definite neurological or psychiatric disorder, including epilepsy or dementia
12. suspected or confirmed history of alcohol or drug abuse;
13. any other condition that, in the opinion of the investigator, makes the patient unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
Piper Fatigue Assessment score | 1 day, 7 days, 14 days, and 28 days postoperatively
  The degree of cancer fatigue was assessed by piper Fatigue Assessment Scale

SECONDARY OUTCOMES:
EORTC QLQ-C30 score | 1 day, 7 days, 14 days, and 28 days postoperatively
  Measure the quality of life of cancer patients in different physical and psychological aspects
EORTC QLQ-BR23 score | 1 day, 7 days, 14 days, and 28 days postoperatively
  Evaluate systemic treatment side effects, arm symptoms, breast symptoms, body image, and sexual function

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Chian/Liaoning, China

IPD SHARING:
Plan to Share IPD: No